CLINICAL TRIAL: NCT06989944
Title: Physical Activity-based Intervention in Depressed Patients: Clinical, Neurophysiological, Epigenetic and Metabolic Correlates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: IRCCS San Raffaele (Other); Istituto Neurologico Mediterraneo Neuromed S. R. L (Other); Azienda Sanitaria Locale di Pescara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PNRR-MCNT2-2023-12377777
Record Dates: First submitted 2025-04-29; First posted 2025-05-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major depressive disorder; physical activity
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA-arm (Experimental): Participants assigned to the PA-arm will participate in at least three weekly 30-minute sessions of PA for a total of 12 weeks.
  Interventions: Behavioral: Physical Activity (PA) program
- Control-arm (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Physical Activity (PA) program — Participants assigned to the PA-arm will participate in at least three weekly 30-minute sessions of PA for a total of 12 weeks.
  The PA program will be tailored to individuals' characteristics, skills and preferences, based on information collected in connection with the baseline assessment and physical examination. A PA program could preview some forms of aerobic/relaxation/anaerobic exercises
  Arms: PA-arm

SUMMARY:
The goal of this clinical trial is to investigate the effect of a structured physical activity (PA) program on depressive symptomatology in adults with a diagnosis of major depression disorder (MDD). The study will evaluate changes in depressive symptoms and assess neurophysiological and biological modulations, including epigenetic, transcriptomic, and metabolic changes resulting from the PA intervention. The main questions it aims to answer are:

* Does physical activity have an impact on depressive symptoms in patients affected by depression?
* What are the neurophysiological, epigenetic, and metabolic mechanisms through which PA can modulate the intensity of depressive symptoms?

Participants will be randomized into two arms: the intervention group (n total=55), in treatment with antidepressants, participating in a 12-weeks PA program; the control group (n total=55), patients in treatment with antidepressants, without receiving the PA program.

All participants will be assessed at three-time points: T0 (baseline, before initiating the trial), T3 (after three months; at the end of the 12-week PA program), and T6 (6th-month follow up; three months after the PA completion).

At each assessment, all participants will:

* Complete clinical evaluation questionnaires
* Provide blood samples
* Undergo electroencephalogram (EEG) measurements.
* Wear an actigraph 24 hours a day for 7 days before the initiation of the trial, at T3, and at T6.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Primary diagnosis of depression (DSM-5 criteria)
* Symptoms of depression according to MADR, BDI, ZDR Scale
* Ability to provide written IC
* Self-reported moderate-intensity leisure PA< 150 min/week

Exclusion Criteria:

* Severe psychopathology
* Medical contraindications to PA (PAR-Q)
* Orthopedic problems/diseases which limit physical fitness assessment
* Currently pregnant (or planning to become pregnant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline (day one), Month 3 (up to three months; end of treatment), Month 6 (up to 6 months; follow up).
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-administered scale designed to assess the severity of depressive symptoms. It consists of 10 items, each rated on a scale from 0 to 6, yielding a total score ranging from 0 to 60. Higher scores indicate greater severity of depression, meaning a worse clinical outcome.
Beck Depression Inventory - II | Baseline (Day 1); Month 3 (up to 3 months; end of treatment); Month 6 (up to 6 months, follow - up)
  The Beck Depression Inventory (BDI) is a self-report questionnaire used to assess the presence and severity of depressive symptoms. It comprises 21 items, each rated on a scale from 0 to 3, resulting in a total score ranging from 0 to 63. Higher scores reflect more severe depressive symptoms, indicating a worse clinical outcome.
Zung Self-Rating Depression Scale | Baseline (Day 1); Month 3 (up to 3 months; end of treatment); Month 6 (up to 6 months, follow - up)
  The Zung Self-Rating Depression Scale (ZDS) is a self-administered questionnaire designed to assess the level of depressive symptoms in individuals. It consists of 20 items, each rated on a scale from 1 to 4, based on how often symptoms are experienced. The raw total score ranges from 20 to 80, which is often converted to an index score (ranging from 25 to 100) by multiplying the raw score by 1.25. Higher scores indicate more severe depression
Personal and Social Performance Scale | Baseline (Day 1); Month 3 (up to 3 months; end of treatment); Month 6 (up to 6 months, follow - up)
  The Personal and Social Performance Scale (PSP) is a clinician-rated instrument used to assess personal and social functioning in individuals with mental disorders. The total score ranges from 1 to 100, with higher scores indicating better functioning and a more favorable clinical outcome.
World Health Organization Quality of Life - Bref | Baseline (Day 1); Month 3 (up to 3 months; end of treatment); Month 6 (up to 6 months, follow - up)
  The WHOQOL-BREF is a self-report questionnaire developed by the WHO to assess quality of life across multiple domains. It contains 26 items rated on a 5-point Likert scale. Higher scores indicate a better quality of life, reflecting a more favorable outcome.

SECONDARY OUTCOMES:
EEG-derived neurophysiological metrics, including spectral, coherence, source localization, and graph-based connectivity measures | Baseline (Day 1); Month 3 (up to 3 months; end of treatment); Month 6 (up to 6 months, follow - up)
  Electroencephalogram (EEG) recordings will be used to derive (a) Individual spectral analysis (theta/alpha transition frequency and individual alpha frequency); (b) Analysis of coherence; c) EEG source localisation with low resolution brain electromagnetic tomograghy; d) Analysis of connectivity.
Metabolic analyses | Baseline (Day 1); Month 3 (up to 3 months; end of treatment)
  Plasma/serum levels of glucose and lipid metabolism markers
Motor activity and circadian/sleep profiles | 24h/day for 7 days before baseline, months 3 (at the end of the trial) and month 6 (up to 6 months follow up)
  Total activity count for every active minute throughout the day wearing an Actigraph accelerometer.
Differentially Expressed genes and biological pathways modulation | Baseline (Day 1); Month 3 (up to 3 months; end of treatment)
DNA Methylation | Baseline (Day 1); Month 3 (up to 3 months; end of treatment)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - IRCCS Centro San Giovanni fi Dio Fatebenefratelli, Brescia
  - Istituto Neurologico Mediterraneo Neuromed, NEUROMED, Isernia
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Sanitaria Locale di Pescara, Pescara